CLINICAL TRIAL: NCT02610920
Title: Identification of Sentinel Lymph Nodes by Ultrasound Utilizing Iron Tracer Injection and Preoperative Biopsy in Women With Breast Cancer
Brief Title: Sentinel Lymph Node Identification in the Axilla of Women With Breast Cancer Using Ultrasound and Iron Injection
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unable to enroll subjects
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAP8967
Record Dates: First submitted 2015-11-15; First posted 2015-11-20 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Breast Neoplasm; Carcinoma, Ductal, Breast; Carcinoma, Intraductal, Noninfiltrating
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast; Carcinoma, Intraductal, Noninfiltrating | interventions — Biopsy; Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Iron-tracer Injection and Biopsy (Experimental): Single injection of 30mg of iron sucrose followed by axillary ultrasound-guided biopsy of lymph node within 2 hours.
  Interventions: Procedure: Iron-tracer guided axillary ultrasound and biopsy; Drug: Iron tracer

INTERVENTIONS:
Procedure: Iron-tracer guided axillary ultrasound and biopsy — After ultrasound identifying sentinel lymph nodes, no more than two nodes will be core-needle biopsied and sent to pathology department for analysis of cancer involvement. The biopsied node(s) will be marked for later identification for the surgeons during the regularly scheduled intraoperative sentinel lymph node biopsy (standard of care).
Drug: Iron tracer — All participants will receive a 30mg injection of subcutaneous iron sucrose into the breast followed by an axillary ultrasound looking for lymph nodes with enhanced reflexivity.
  Other Names: Venofer; 75010550

SUMMARY:
This study evaluates a new method of testing the lymph nodes in the armpit of patients with breast cancer for tumor involvement. All participants involved in this study will undergo an injection of a small amount of iron dissolved in liquid followed by an ultrasound of the axilla that will make previously invisible lymph nodes visible, allowing them to be sampled in an outpatient setting.

DETAILED DESCRIPTION:
Lymph nodes are small collections of tissue all over the body that drain bodily fluid. These axillary lymph nodes are important in evaluating breast cancer since, if they are positive, it suggests that the cancer cells have spread outside of the breast. The current standard of care is for most breast cancer patients undergoing surgery to have a sentinel lymph node biopsy which is a procedure to take a sample of the lymph nodes in the armpit (also called the axilla) during their breast surgery. However this intraoperative biopsy comes with certain risks such as arm swelling or lymphedema, arm pain, arm numbness/tingling, and/or psychological distress from waiting for the results or the possibility of further interventions. In order to avoid this and have a result before surgery, this study will explore a nonsurgical method of sampling these lymph nodes. Normally suspicious lymph nodes are hard to find accurately by exam and ultrasound.

A new method has been developed that involves injecting a small amount of iron dissolved in liquid into the breast that gets absorbed by the lymph nodes making them bright on ultrasound and possible to biopsy. This method has been shown to have results as accurate as standard sentinel lymph node biopsy by comparing them in the operating room. This study will now investigate performing these ultrasounds and biopsies in the office as well as compare these results to the results of the standard sentinel lymph node biopsy in the operating room. The results of this study could help future breast cancer patients to avoid invasive sampling and all of the accompanying risk as well as give patients and the care team an idea of the extent of disease sooner in order to guide management.

ELIGIBILITY:
Inclusion Criteria:

* Female patients at least 21 years old
* Patients with invasive ductal carcinoma staged T1 or T2 with estrogen receptor and progesterone receptor positive (ER+/PR+) who are scheduled for sentinel lymph node biopsy
* Patients with Ductal Carcinoma In Situ (DCIS) (high or low grade) who are scheduled for sentinel lymph node biopsy including:
* Patients having a mastectomy
* Patients with palpable DCIS
* Patients undergoing breast conservation with large (>5cm) area of DCIS
* Patients with signed consent to participate

Exclusion Criteria:

* Preoperative palpable axillary lymphadenopathy
* Preoperative ultrasound demonstrating suspicious adenopathy
* Previous axillary dissection or previous lymph node biopsy
* Patients with Invasive Lobular Carcinoma
* Patients who are pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12 (Estimated); Primary Completion 2017-06 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of core needle biopsy of sentinel lymph node | At time of surgery, about 7 days after initial core needle biopsy
  The participants will undergo an outpatient iron tracer-guided ultrasound and axillary lymph node core needle biopsy at "day zero" (purposely done no more than 7 days prior to scheduled breast surgery). The investigators would like to see if this biopsied node was in fact the sentinel lymph node. This will be determined by all of the patients also undergoing their previously scheduled intraoperative sentinel lymph node biopsy (standard of care) at about day 7. The success rate will measure what percentage of the preoperative lymph nodes biopsied with this novel technique were truly sentinel lymph node(s).

SECONDARY OUTCOMES:
Concordance rate of core needle biopsy pathology to sentinel lymph node biopsy pathology | At time of pathology reports, about 17 days after initial core needle biopsy
  The investigators will measure the concordance rate of the novel iron-tracer guided lymph node core needle biopsy pathology results (determining if cancer cells are present or not) compared to the operative sentinel lymph node pathology results. The novel technique core needle biopsy will occur on day zero. The surgery with concurrent sentinel lymph node biopsy will be on or before day 7, and both pathology reports should be back by day 17.

CONTACTS AND LOCATIONS:
Overall Officials: Bret Taback, MD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kusminsky RE, Witsberger T, Todd Kuenstner J, Willis Trammell S, Schlarb CA, Maxwell D, Richmond BK, Boland JP. Identification of the sentinel node by ultrasonography in patients with breast cancer. Ann Surg Oncol. 2014 Jun;21(6):1969-74. doi: 10.1245/s10434-014-3570-4. Epub 2014 Feb 25. PMID 24566860
- [Background] Bailie GR. Comparison of rates of reported adverse events associated with i.v. iron products in the United States. Am J Health Syst Pharm. 2012 Feb 15;69(4):310-20. doi: 10.2146/ajhp110262. PMID 22302256